CLINICAL TRIAL: NCT06601296
Title: STING Agonist and Personalized Ultra-fractionated Stereotactic Adaptive Radiotherapy in Combination With Checkpoint Inhibition for Patients With Metastatic Kidney Cancer.
Brief Title: Radiotherapy in Combination With Checkpoint Inhibition for Patients With Metastatic Kidney Cancer
Acronym: SPARK
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Raquibul Hannan, MD, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0919
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Renal Cell Carcinoma ( mRCC); OligoProgressive Metastatic Disease
Keywords: renal; kidney; mrcc; metastatic; cancer; STING; PULSAR; SABr; SPARK; nivolumab; IMSA 101
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis; Neoplasms; Bites and Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SAbR with Intratumoral STING agonist IMSA101 and IO with Anti-PD1 (Experimental): Only one arm will be maintained in this phase II study with all patients undergoing the following treatment:
  SOC treatment: Nivolumab 480 mg monthly PULSAR: 36 Gy in 3 fractions, Q4weeks IMSA101: three intra-tumoral injections of one of the progressive lesions at 1200 mcg (C1D1, C2D1, C3D1)
  Interventions: Drug: IMSA101

INTERVENTIONS:
Drug: IMSA101 — All enrolled patients to undergo the following treatment:
  SOC treatment: Nivolumab 480mg monthly PULSAR: 36 Gy in 3 fractions, Q4weeks IMSA101: three intra-tumoral injections of one of the progressive lesions at 1200 mcg (C1D1, C2D1, C3D1)

SUMMARY:
To evaluate the impact of combining innate immune system activation (with IMSA101) with antigen release (through SAbR/PULSAR) on limited progressing lesions during ongoing adaptive immune system activation (with maintenance Nivo).

DETAILED DESCRIPTION:
The study expects to accrue the 15 patients over a 3-4 year period.

Patients with oligoprogressive disease (≤5 lesions) after treatment with Anti-PD1 / Anti-CTLA-4 will continue Anti-PD1 (nivolumab). All patients will have a mandatory PD-L1 PET (Pre-treatment and Week 12). All patients will undergo baseline biopsy (just before the administration of IMSA101 of the same lesion to be injected). SAbR will be delivered in 3 fractions at 12 Gy every 4 weeks (PULSAR regimen) to all progressing lesions. One lesion will also receive 3 intratumoral injections of IMSA101 (C1D1, C1D8, C1D15, C2D1, C3D1) immediately after radiation either on the same day or within 72 hours after the PULSE.

Selected Phase 2 dosing of IMSA101 (1200mcg) will be utilized.

At disease progression, patients have the option to undergo additional imaging and tissue/blood collections.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have metastatic ccRCC.
* Patients must have oligoprogression defined as progression in ≤5 lesions.
* All oligoprogression lesions must be suitable for radiation.
* Patients must have at least one site of disease that can be safely injected with IMSA101.
* Karnofsky Performance Status (KPS) of at least 50%.
* Age ≥ 18 years.
* Patients must have adequate organ and marrow function within 14 days prior to study entry.
* All IMDC risk categories are allowed.

Exclusion Criteria:

* Patients with progressive ultracentral/central chest lesions will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate the PFS rate associated with the therapeutic intervention. PFS is defined as the duration of time from initiation of PULSAR/IMSA101 to disease progression as defined by RECIST1.1 or death. | Time from initiation of PULSAR/IMSA101 until death from any cause. Follow-up visits to be done every 12 weeks (+/- 1 week) for study duration until patient has progressed. Afterward, subjects to be contacted every 6 months for survival data up to 5 years
  Exact binomial test will be used to test if the lower limit of the 95% confidence interval of the probability of postponing systemic therapy >9 months will be greater than 30%.

CONTACTS AND LOCATIONS:
Overall Officials: RAQUIBUL HANNAN, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States